CLINICAL TRIAL: NCT04904848
Title: Cultural Adaptation, Validity and Reliability of the Turkish Version of the "Children's Assessment of Participation With Hands (CAP-H)" Scale in Children With Physical Disabilities
Brief Title: Turkish Version of the "Children's Assessment of Participation With Hands Scale
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin,PT, Principal Investigator, Pamukkale University
Other Study IDs: 2019-192
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Participation, Patient; Child, Only
Keywords: validity; reliability; children; participation; hand
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey evaluation — examine the convergent validity and reliability of a Turkish version

SUMMARY:
To the best of our knowledge, there is no Turkish validity and reliability scale that can reveal children's hand involvement. In the study in which the CAP-H was developed, it was stated that this scale could be used in population-level research studies to examine the similarities and differences in children's manual life participation among different diagnosis groups. It is very important to adapt translated assessment tools to different cultures and languages and to verify their reliability and validity. Moreover, self-report questionnaires are advantageous in that they can be used for large-scale testing. The aim of this study was to examine the convergent validity and reliability of a Turkish version of the "Children's Assessment of Participation with Hands (CAP-H)" scale in order to evaluate the hand participation of physically disabled children.

DETAILED DESCRIPTION:
The CAP-H scale was used to evaluate children's hand participation and to examine the validity and reliability of the Turkish version. The original scale was developed by Chien et al. in Australia in 2015 to evaluate the difficulties experienced by children aged 2-12 years in using the hands in daily living activities that require hand participation. In the adaptation of the CAP-H to Turkish, the standard protocol of the WHO for the adaptation of the scales to different languages was applied:

1. Translation of the scale into the target language (forward translation)
2. Review of the scale translated into the target language by an expert panel of 2 pediatric rehabilitation physiotherapists, who can speak both languages.
3. Translation of the scale from the target language to the original language (back translation)
4. Testing the translated scale and discussing its conceptual integrity
5. Final version of the adapted scale (final version)

For validity of CAP-H, Gross Motor Function Classification System and Manual Assesment Classification System scales used.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation in the study,
* having a physical disability report,
* the evaluated child in the age range of 2-12 years, and
* the respondent (child or parent) to be Turkish literate

Exclusion Criteria:

* Do not want to participate in the study
* Not completing surveys

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with physical disability
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Children's Assessment of Participation with Hands (CAP-H)" scale | 2 week
  The original scale was developed by Chien et al. in 2015 to evaluate the difficulties experienced by children aged 2-12 years in using the hands in daily living activities that require hand participation. The scale consists of 32 items in 4 sections: self-care participation (9 items), recreational participation (11 items), educational participation (8 items), and domestic life and community participation (9 items). Each section has 4 sub-scores of difference, frequency, independence and desire to change sections, scored with Likert-type responses, and higher scores indicate higher hand participation. The percentage score is obtained by dividing the total score by the number of items marked in the sub-scores of difference and change request. In frequency and independence scoring, the score is obtained by dividing the total score by the number of items marked.

SECONDARY OUTCOMES:
Gross Motor Function Classification System | 1 week
  The (GMFCS), developed for children, is a classification system based on the child's self-initiated movements with an emphasis on sitting, displacement and mobility. Since the motor functions of children vary depending on age, functions for each age group are defined for each level, including children under 2 years old, between 2 and 4 years old, between 4 and 6 years old, and between 6 and 12 years old. While it was previously used for children under the age of 12 years, it can now be used for young people between the ages of 12 and 18 years in its expanded form.
  GMFCS levels according to age Level I: walks without restrictions Level II: Walks with restrictions Level III: Walks using hand-held mobility aids Level IV: Self-movement is restricted; can use motor mobility vehicle. Level V: Transported in a hand-pushed wheelchair
Manual Assesment Classification System | 1 week
  The Manual Assesment Classification System (MACS) is used to classify children's ability to hold objects in daily activities. Turkish validity and reliability studies have been conducted. While MACS evaluates the participation of both hands together in activities, it cannot evaluate the hands separately. The classification is graded as follows:
  I - Holds objects easily and successfully. II- Can hold many objects, but the speed and / or quality of achievement is somewhat reduced.
  III- Holds objects with difficulty; help is needed in modifying and / or organizing activities.
  IV- Holds a selected limited number of objects easily arranged in adapted situations.
  V- Cannot hold objects and has severely limited ability to perform even a simple action.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Yaprak Cetin, Assoc, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will share our data with other researchers by Statistical Package Program

REFERENCES:
- [Result] Chien CW, Rodger S, Copley J. Development and Psychometric Evaluation of a New Measure for Children's Participation in Hand-Use Life Situations. Arch Phys Med Rehabil. 2015 Jun;96(6):1045-55. doi: 10.1016/j.apmr.2014.11.013. Epub 2014 Nov 29. PMID 25437107
- Available data/document: Individual Participant Data Set — http://pubmed.ncbi.nlm.nih.gov/25437107/